CLINICAL TRIAL: NCT01105286
Title: A Psoriasis Plaque Test Comparing Eight Different Formulations of Vitamin D Analogues for the Treatment of Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PLQ-005; 2009-017393-20 (EudraCT Number)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-10

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcipotriol ointment (Experimental)
  Interventions: Drug: Six different calcipotriol ointment formulations, and two currently marketed topical vitamin D analogues

INTERVENTIONS:
Drug: Six different calcipotriol ointment formulations, and two currently marketed topical vitamin D analogues — Once daily application

SUMMARY:
The purpose of this trial is to compare the anti-psoriatic effect of eight different formulations of vitamin D analogues using a psoriasis plaque test design

ELIGIBILITY:
Inclusion Criteria:

* Subjects having understood and signed an informed consent form.
* Either sex
* Age 18 years or above
* All skin types and any ethnic origin
* Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs or trunk.

Exclusion Criteria:

* Females who are pregnant, or who wish to become pregnant during the study, or who are breast feeding
* Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks/5 half-lives (which-ever is longer) for experimental biological products prior to randomisation
* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immuno-suppressants) within the 4-week period prior to randomisation
* Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation and during the study:

  * Potent or very potent (WHO group III-IV) corticosteroids
  * PUVA or Grenz ray therapy
* Subjects using one of the following topical drugs for the treatment of psoriasis within two weeks prior to randomisation and during the study:

  * WHO group I-II corticosteroids (except if used for treatment of scalp psoriasis)
  * Topical retinoids
  * Vitamin D analogues
  * Topical immunomodulators (e.g. macrolides)
  * Anthracen derivatives
  * Tar
  * Salicylic acid
  * UVB therapy
* Subjects known to be non-responder to topical vitamin D analogues (e.g., known history of no improvement or worsening of psoriasis with e.g., calcipotriol, calcitriol or tacalcitol when used according to current SmPc)
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments)
* Subjects with current participation in any other interventional clinical, based on interview of the subject
* Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
* Subjects with known or suspected hypersensitivity to component(s) of the investigational products
* Subjects with known/suspected disorders of calcium metabolism associated with hypercalcaemia
* Subjects with known severe hepatic and/or severe renal insufficiency
* Subjects with any concomitant medical or dermatological disorder(s) which might preclude accurate evaluation of the psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Total Clinical Score of clinical symptoms | 4 weeks

SECONDARY OUTCOMES:
Clinical scores, lesions thickness | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Facy, PhD, Study Director — LEO Pharma
Locations (1):
- LEO Pharma investigational site, Nice, France

IPD SHARING:
Plan to Share IPD: No